CLINICAL TRIAL: NCT01270217
Title: Behavior and Driving Safety Study II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Sacramento Police Department (Unknown); California Office of Traffic Safety (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201018332
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Alcoholic Intoxication
Keywords: Automobile driving; Driving under the influence; Interview, psychological; Brief intervention; Brief motivational interview
MeSH Terms: conditions — Alcoholic Intoxication; Driving Under the Influence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief motivational interview (Experimental)
  Interventions: Behavioral: Brief motivational interview
- No discussion (No Intervention)

INTERVENTIONS:
Behavioral: Brief motivational interview — The brief motivational interview is a non-confrontational, patient-centered discussion between a counselor (e.g., social worker, nurse, physician, or psychologist) and an at-risk individual during which the individual's motivation and confidence to change health-related behaviors are explored.
  Arms: Brief motivational interview

SUMMARY:
The purpose of this study is to determine whether brief motivational interviews reduce problematic drinking behavior among individuals arrested for the first time for driving under the influence of alcohol (DUI).

DETAILED DESCRIPTION:
Despite extensive legislative, law enforcement, and public awareness efforts, driving under the influence of alcohol (DUI) remains a major cause of mortality and loss of years of productive life. A brief motivational interview (BI) is a non-confrontational, patient-centered discussion during which the individual's motivation and confidence to change health-related behaviors are explored. Previous studies of BIs in health care settings suggest that BIs administered after hospitalization for alcohol-related injury reduce the likelihood of repeat injury hospitalization and arrest for DUI. This study will evaluate whether brief motivational interviews reduce problematic drinking behavior among individuals arrested for the first time for driving under the influence of alcohol (DUI).

ELIGIBILITY:
Inclusion Criteria:

* First arrest for driving under the influence of alcohol
* Arrest involved operation of a motor vehicle
* At least 18 years of age
* English-speaking

Exclusion Criteria:

* Arrest involved injury to another person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test score | 3 months

SECONDARY OUTCOMES:
Time to repeat arrest for driving under the influence of alcohol | Up until one year after the conclusion of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Garth H Utter, MD MSc, Principal Investigator — University of California, Davis
Locations (1):
- Sacramento County Main Jail, Sacramento, California, United States

REFERENCES:
- [Derived] Utter GH, Young JB, Theard LA, Cropp DM, Mohar CJ, Eisenberg D, Schermer CR, Owens LJ. The effect on problematic drinking behavior of a brief motivational interview shortly after a first arrest for driving under the influence of alcohol: a randomized trial. J Trauma Acute Care Surg. 2014 Mar;76(3):661-70; discussion 670-1. doi: 10.1097/TA.0000000000000144. PMID 24553532